CLINICAL TRIAL: NCT02631265
Title: Reduction of Basal Insulin to Prevent Hypoglycemia During Exercise in Adults With Type 1 Diabetes Using Insulin Pump Therapy
Brief Title: Insulin-based Strategies to Prevent Hypoglycemia During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Professor of medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RIDE-1
Record Dates: First submitted 2015-12-10; First posted 2015-12-16 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Exercise; Hypoglycemia; Insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reduction of insulin basal rate at the time of exercise (Active Comparator)
  Interventions: Other: Exercise 1
- Reduction of insulin basal rate 20 minutes prior to exercise (Active Comparator)
  Interventions: Other: Exercise 2
- Reduction of insulin basal rate 40 minutes prior to exercise (Active Comparator)
  Interventions: Other: Exercise 3

INTERVENTIONS:
Other: Exercise 1 — Participants will be admitted at IRCM at 14:00. At 15:30, participant's insulin basal rate will be reduced by 80% and participants will perform a 45-minute exercise on the ergocycle at 60% of VO2 peak (moderate intensity). At 16:15, the participant's usual insulin basal rate will be set in the insulin pump and a standardized snack (30g CHO) will be served. At 16:45, the participant will be discharged and will be asked to eat a standardized dinner at home (60g CHO for females and 80g CHO for males).
  Arms: Reduction of insulin basal rate at the time of exercise
Other: Exercise 2 — Participants will be admitted at IRCM at 14:00. At 15:10, participant's insulin basal rate will be reduced by 80%. At 15:30, participants will perform a 45-minute exercise on the ergocycle at 60% of VO2 peak (moderate intensity). At 16:15, the participant's usual insulin basal rate will be set in the insulin pump and a standardized snack (30g CHO) will be served. At 16:45, the participant will be discharged and will be asked to eat a standardized dinner at home (60g CHO for females and 80g CHO for males).
  Arms: Reduction of insulin basal rate 20 minutes prior to exercise
Other: Exercise 3 — Participants will be admitted at IRCM at 14:00. At 14:50, participant's insulin basal rate will be reduced by 80%. At 15:30, participants will perform a 45-minute exercise on the ergocycle at 60% of VO2 peak (moderate intensity). At 16:15, the participant's usual insulin basal rate will be set in the insulin pump and a standardized snack (30g CHO) will be served. At 16:45, the participant will be discharged and will be asked to eat a standardized dinner at home (60g CHO for females and 80g CHO for males).
  Arms: Reduction of insulin basal rate 40 minutes prior to exercise

SUMMARY:
It has been reported that insulin basal rate reduction initiated at exercise onset can reduce the hypoglycemic risk during exercise. However, another potentially more efficient strategy to prevent exercise-induced hypoglycemia could be to reduce insulin basal rate a certain time prior to exercise. No study investigated what would be the best timing to initiate such temporary basal insulin reduction. Therefore, the objective of this study will be to compare the efficacy of three strategies to prevent exercise-induced hypoglycemia during a 45 min exercise at 60% VO2peak (moderate intensity): 1) reduce insulin basal rate at the time of exercise; 2) reduce insulin basal rate 20 minutes prior to exercise; 3) reduce insulin basal rate 40 minutes prior to exercise. Investigators hypothesize that the time spent in hypoglycemia will be less when the insulin basal rate is reduced 40 minutes prior to exercise compared to a reduction at the time of exercise. Secondary hypotheses are: 1) Time spent in hypoglycemia will be less when the insulin basal rate is reduced 20 minutes prior to exercise compared to a reduction at the time of exercise; 2) Time spent in hypoglycemia will be less when the insulin basal rate is reduced 40 minutes prior to exercise compared to a reduction 20 minutes prior to exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. The subject will have been on insulin pump therapy for at least 3 months.
4. Last (less than 2 months) HbA1c ≤ 12%.

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy (especially diagnosed gastroparesis) or severe proliferative retinopathy as judged by the investigator.
2. Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Abnormal blood panel and/or anemia.
4. Ongoing pregnancy.
5. Severe hypoglycemic episode within two weeks of screening.
6. Other serious medical illness likely to interfere with study participation or with the ability to complete the exercise periods by the judgment of the investigator (e.g. orthopedic limitation).
7. Failure to comply with team's recommendations (e.g. not willing to change pump parameters, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Percentage of time of capillary blood glucose levels spent below 4 mmol/L | This outcome will be measured over 45 minutes.
  This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15

SECONDARY OUTCOMES:
Decrease in glucose levels | This outcome will be measured over 45 minutes.
  Difference between glucose levels at the beginning of the exercise and the lowest glucose level from the start of the exercise until the end of exercise. This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15
Decremental area under the curve of sensor glucose levels | This outcome will be measured over 45 minutes.
  This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15
Area under the curve of sensor glucose levels < 4 mmol/L | This outcome will be measured over 45 minutes.
  This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15
Number of patients with an exercise-induced hypoglycemia < 3.9 mmol/L | This outcome will be measured over 45 minutes.
  This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15
Number of patients with an exercise-induced hypoglycemia < 3.5 mmol/L | This outcome will be measured over 45 minutes.
  This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15
Number of patients requiring an oral treatment for hypoglycemia | This outcome will be measured over 45 minutes.
  This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15
Total number of hypoglycemia episode requiring treatment | This outcome will be measured over 45 minutes.
  This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15
Percentage of time spent between 4 and 10 mmol/L | This outcome will be measured over 45 minutes.
  This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15
Mean time (minutes) to the first hypoglycemic event | This outcome will be measured over 45 minutes.
  This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15
Percentage of time spent < 4.0 mmol/L | This outcome will be measured over 14.75 hours.
  This time frame corresponds to the post-exercise period, from the end of the exercise until 7:00 the next morning.
Percentage of time of sensor glucose levels spent below 4 mmol/L | This outcome will be measure over 45 minutes
  This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15
Absolute difference between capillary blood glucose levels and sensor glucose levels | This outcome will be measure over 45 minutes
  This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15
Relative difference between capillary blood glucose levels and sensor glucose levels | This outcome will be measure over 45 minutes
  This time frame corresponds to the exercise period. The exercise period will be from 15:30 to 16:15

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No